CLINICAL TRIAL: NCT02828332
Title: Study of Developmental Trajectories From Childhood to Adulthood Patients of the Cohort EpiTED: Research for Prognostic Factors Clinical and Biological
Brief Title: Developmental Trajectories in ASD Until Adulthood: A 15 Years Follow-up Study
Acronym: EpiTED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 8878
Record Dates: First submitted 2016-07-05; First posted 2016-07-11 (Estimated); Last update posted 2016-07-11 (Estimated); Status verified 2016-03

CONDITIONS: Autism Spectrum Disorders
Keywords: Autism Spectrum Disorders; Cohort
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Quality of Life

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patient with autism disorder (Other): Interview with a psychologist who do Vineland II (VABS -II) and evaluate Quality of life and comorbidities
  Interventions: Other: Vineland II (VABS -II); Other: Quality of life

INTERVENTIONS:
Other: Vineland II (VABS -II) — semi-structured interview with a psychologist; Measure 4 areas: Communication, skills of daily living, socialization and skills Motrices
Other: Quality of life — Evaluation of the quality of life and comorbidities

SUMMARY:
Epidemiological studies have shown that a wide range of outcome trajectories exist in ASD, but little is known about their determinant in a long-term perspective. The EpiTED cohort was set-up in order to understand the heterogeneity of developmental trajectories among children with a diagnosis of PDD and the role of clinical, biological and environmental factors in their adaptive outcome. It is one of the rare cohorts involving a long term prospective follow-up based on a large set of variables, and precise phenotypes of the entire autism spectrum.

DETAILED DESCRIPTION:
Purpose: Epidemiological studies have shown that a wide range of outcome trajectories exist in ASD, but little is known about their determinant in a long-term perspective. The EpiTED cohort was set-up in order to understand the heterogeneity of developmental trajectories among children with a diagnosis of PDD and the role of clinical, biological and environmental factors in their adaptive outcome. It is one of the rare cohorts involving a long term prospective follow-up based on a large set of variables, and precise phenotypes of the entire autism spectrum.

Participants: This longitudinal study for which recruitment began between 1997 and 1999, has initially involved 281 preschool aged children recruited from 5 French areas. They were seen at 8 (Time 2), 15 (Time 3) and 20 years of age (Time 4), with an average follow-up length of 15 years. At each follow-up, socio-demographical, clinical, developmental and interventional were collected. At Time 4 (fourth visit), DNA was collected to do a genetic study Findings to date: The main results show that there were two developmental trajectories from childhood to adolescence among the cohort leading to very distinct level of adaptive functioning. Prognosis factors in childhood were the intellectual level, the presence or absence of language, the autism degree and the absence or presence of epilepsy. During adolescence there was a negative impact on the quality of life of the parents of the presence of aberrant behavior and low level functioning, The children included in the cohort were followed during 15 years and were assessed four times (at 5, 8, 15 and 20 years on average, see flow chart in figure 1. From 2000 to 2002, 219 of the original group were reassessed (time 2, T2). At time 3 (T3), between 2007 and 2009, they were 152 to be re-assessed and 106 between 2012 and 2015 (time 4, T4).

ELIGIBILITY:
Inclusion Criteria:

* Patients previously include in the troop constituted in 1997 /1999 as part of PHRC 96/97 and having been followed during 10 years.
* Patients are 18
* Patients with diagnosis of infantile autism or atypical autism according to the criteria of the CIM 10 at the time of their initial inclusion.

Exclusion Criteria:

* Refusal of participation
* Women pregnant breastfeeding
* persons deprived of freedom by court order

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2012-10; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Vineland II (VABS -II) | 1 day
  semi-structured interview with a psychologist; Measure 4 areas: Communication, skills of daily living, socialization and skills Motrices

SECONDARY OUTCOMES:
Quality of life | 1 day
  Evaluation of quality of life by questionnaire
comorbidities | 1 day
  Evaluation comorbidities by a clinician directed interview

CONTACTS AND LOCATIONS:
Overall Officials: Amaria Baghdadli, MCU-PH, Principal Investigator — CHU de Montpellier

IPD SHARING:
Plan to Share IPD: No